CLINICAL TRIAL: NCT05739591
Title: Registry for Long-term Follow-up of Safety and Efficacy Parameters of GBG Study Participants
Brief Title: Long-term Safety and Efficacy of GBG Study Participants
Acronym: ETERNITY
Status: Recruiting | Type: Observational
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: GBG 107
Record Dates: First submitted 2023-02-05; First posted 2023-02-22 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Registry; Breast cancer, early; Safety; Efficacy; Long-term follow-up; Long-term survival; German Breast Group
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — In case of distant disease recurrence, it is recommended - according to guidelines - to confirm diagnosis by histological examination of the metastatic lesion. By signing the informed consent form, the patient agrees to the transfer of biomaterial to GBG.
  If a histological examination of a metastasis was performed by standard of care, a formalin-fixed paraffin-embedded (FFPE) tumor tissue block from the metastatic lesion should be provided to GBG. Method of material collection (i.e., diagnostic biopsy or surgery) is not part of the registry.
  The submitted tumor samples will be used for translational research objectives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ETERNITY study is an international, multicenter, observational study that aims to follow up patients who have participated in a GBG trial for early breast cancer, even after the study has officially ended, in order to collect long-term data on survival, late or delayed adverse events, in addition to information related to pregnancy, fertility and other parameters impacting quality of life.

DETAILED DESCRIPTION:
This is a prospective and retrospective, international, multicenter, non-interventional, observational study for collection of long-term safety and efficacy parameters of former GBG study participants of prospective clinical trials on early breast cancer.

Patients with prospective data collection will be informed about the registry by the treating physician at the study site. After written informed consent (which may already be included in the main and/or biomaterial informed consent form of the respective clinical study) for data and biomaterial collection, the registration form will be filled out completely within the GBG electronic data capture system (MEDCODES®). Inclusion and registration can take place after informed consent of the patient. However, documentation of follow-up should start after the regular end of study or with the start of the follow-up period, as defined in the respective study protocol.

A correlation of the follow-up registry database with the respective study databases is possible via the patient identification number of the participant. Consequently, the long-term effects of the study therapy can be calculated per therapy group, and the effectiveness can be correlated with possible late-onset toxicities.

Post-study long-term outcome follow-up will be assessed according to local/national guidelines for standard follow-up examinations and post-treatment surveillance. Data should be documented at least once a year in the registry.

Relapse and safety assessment will be performed, and survival status will be collected in all registered patients. Here, the investigator may conduct evaluations or assessments within regular follow-up visits. However, telephone contact or contact in writing with the patient or treating physician or relatives in case of death is also acceptable. Imaging tests (e.g., mammography and/or staging workup) are recommended according to local/national guidelines for follow-up and in case of symptoms suspicious for locoregional or distant relapse.

Information to be collected include:

* Date and site of first non-invasive local recurrence, first invasive local recurrence, first contralateral breast recurrence, first regional recurrence, first distant recurrence
* Date and diagnosis of secondary malignancies
* Date and cause of deaths
* Pregnancies after study participation and their respective outcome
* Anti-hormonal therapies in HR+ breast cancer patients
* Further anti-cancer treatments after study participation
* Long-term adverse drug reactions of the respective study treatments

In case of disease recurrence, it is recommended to confirm diagnosis by histological examination. If performed, an FFPE tumor tissue block from the metastatic lesion should be provided to GBG.

It is allowed and recommended to register patients in parallel in the GBG self-reporting registry (available only in German) that will allow follow-up and long-term efficacy evaluations beyond the end of the respective study by the patients themselves.

STATISTICS

This is an observational study for collection of long-term safety and efficacy parameters of former GBG study participants. As long-term outcomes and late-onset toxicities are also secondary objectives in all prospective clinical studies of the GBG, statistical methods will adhere as much as possible to methods described in the respective clinical trial protocols.

For the analysis, data from the corresponding clinical trials (e.g., baseline characteristics, short-time efficacy, and toxicity parameters, already collected follow-up data, etc.) will be merged with the registry data.

DATA HANDLING, MANAGEMENT AND QUALITY ASSURANCE

The GBG EDC system MEDCODES® will be maintained by GBG Forschungs GmbH for all study sites.

Data management, which comprises CRF design, database and application hosting, data entry, and data validation, will be performed by GBG Forschungs GmbH for all study sites. GBG Forschungs GmbH will provide the investigator site with the web base EDC system MEDCODES® that is validated and conforms to 21 CFR Part 11 requirements. Investigator site staff will not be given access to MEDCODES® until they have been trained on the EDC system.

Visual and computerized methods of data validation are applied in order to ensure accurate, consistent, and reliable data for the subsequent analyses.

All communication between MedCODES® and the clients is securely encrypted (Secure HTTP).

In order to protect patient confidentiality, each participating patient is assigned a unique GBG patient identification number. Instead of the true patient identity, the pseudonym is used in all communication between the trial site and the GBG Forschungs GmbH. A correlation of the follow-up registry database with the respective study databases is possible via the patient identification number of the participant.

Every user is provided with a unique username and a unique password. Every user is assigned to a user group which represents their role in the CRF workflow. Access control is based on user name, group. Therefore, users can only access those datasets necessary for them to fulfill their role in the CRF workflow ("need to know basis").

ELIGIBILITY:
Inclusion criteria:

* Participation and treatment in a GBG clinical trial for early breast cancer.
* Prospective registration: Written informed consent according to local regulatory requirements prior to data and biomaterial collection.

Exclusion criteria:

* Participation and treatment in a non-GBG clinical trial for early breast cancer.
* Patients with advanced or metastatic breast cancer who have participated and received treatment in a GBG clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated and received treatment as part of a GBG clinical trial for early breast cancer.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2030-05-19 (Estimated); Study Completion 2030-05-19 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 10 years
  Time period between randomization and first event (ipsi- or contralateral (non-) in-breast or loco-regional recurrence, distant recurrence, death from breast cancer, death from non-breast cancer cause, death from unknown cause, invasive contralateral breast cancer, second primary invasive cancer (non-breast))
Invasive disease-free survival (iDFS) | 10 years
  Time period between randomization and first event (ipsi- or contralateral invasive in-breast or loco-regional recurrence, distant recurrence, death from breast cancer, death from non-breast cancer cause, death from unknown cause, invasive contralateral breast cancer, second primary invasive cancer (non-breast))
Distant disease-free survival (DDFS) | 10 years
  Time period between randomization and diagnosis of any distant recurrence of disease, any second primary invasive cancer (non-breast) or death due to any cause, whichever occurs first
Locoregional recurrence-free survival (LRRFS) | 10 years
  Time period between randomization and diagnosis of any loco-regional (ipsilateral breast (invasive or DCIS), local/regional lymph nodes) recurrence of disease, any invasive contralateral breast cancer or death due to any cause, whichever occurs first
Overall survival (OS) | 10 years
  Time period between randomization and death of any cause
Other primary outcome measures | 10 years
  Other study-specific long-term survival endpoints may be defined in the respective study protocol or statistical analysis plan (SAP)

SECONDARY OUTCOMES:
Long-term toxicity | 10 years
  Frequency and severity of long-term toxicity associated with study treatment are graded by the current NCI Common Terminology Criteria for Adverse Events version (NCI-CTCAE) or according to the respective study protocol or statistical analysis plan (SAP)
Anti-cancer therapies | 10 years
  Anti-cancer therapies including anti-hormonal therapy in hormone receptor positive (HR+) breast cancer after study participation are analyzed descriptively
Pregnancies | 10 years
  Pregnancies after study participation and their outcome are analyzed descriptively.
Impact of study treatment on Quality of Life (QoL) | 10 years
  In this registry, two questions on content on quality of life and degree of bother by side-effects are used

OTHER OUTCOMES:
Explorative translational research endpoints | 10 years
  Correlation of explorative biomarkers with survival and toxicity endpoints. Details are defined in the corresponding SAP

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Loibl, Prof. Dr., Study Chair — GBG Forschungs GmbH
Locations (3):
- Austria (3):
  - MUI - Univ. Klinik f. Frauenheilkunde Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH - BHS, Linz
  - LKH Salzburg - PMU, Salzburg